CLINICAL TRIAL: NCT03323242
Title: -SEALIVE- The Use of Technical Vessel Sealing Devices for Recipient Hepatectomy in Liver Transplantation: Study Protocol for a Randomized Controlled Trial
Brief Title: The Use of Technical Vessel Sealing Devices for Recipient Hepatectomy in Liver Transplantation
Acronym: SEALIVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. A. Mehrabi, MD, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-217/2017
Record Dates: First submitted 2017-09-07; First posted 2017-10-26 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Hepatectomy
Keywords: Vessel Sealing Devices; Liver Transplantation

STUDY DESIGN:
Masking Description: Blinding the surgical staff is impossible due to the use of different methods in the three groups under investigation. Since the primary endpoint "total blood loss" will be precisely recorded during surgery by independent staff and secondary endpoints are objective physiological findings, blinding the subjects is not needed. Therefore, the open design is not expected to cause any avoidable bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Recipient hepatectomy using conventional bipolar coagulation devices, surgical suture ligatures, and surgical clips (or any dissecting / coagulating device other than LS)
- LS group (Experimental): Recipient hepatectomy applying LigaSure.
  Interventions: Device: LigaSure
- USD group (Experimental): Recipient hepatectomy applying Harmonic Ultrasonic dissector.
  Interventions: Device: Harmonic Ultrasonic dissector

INTERVENTIONS:
Device: LigaSure — The dissection of the small blood vessels and the connective tissue in the hepatoduodenal ligament is carried out with LigaSure
  Arms: LS group
Device: Harmonic Ultrasonic dissector — The dissection of the small blood vessels and the connective tissue in the hepatoduodenal ligament is carried out with Harmonic Ultrasonic dissector
  Arms: USD group

SUMMARY:
The surgical technique used in liver transplantation has undergone constant Evolution in an effort towards towards a safe, highly standardized procedure. Despite this, the initial step of the recipients' hepatectomy has not been in the focus of clinical research thus far. Due to usually advanced coagulopathy in liver transplantation recipients, this part of the operation still bares the risk of severe hemorrhage. This trial is designed to compare an electrothermic, bipolar vessel sealing device (LigaSureTM) and an ultrasound dissector (HARMONIC ACE®+7) to standard surgical techniques during the recipients' hepatectomy in liver transplantation. In a single center, prospective, randomized, controlled, parallel three armed, confirmatory, open trial, LigaSureTM and HARMONIC ACE®+7 will be compared to standard surgical techniques which, utilize titanium clips and conventional knot tying ligations during the recipients' hepatectomy in liver transplantation. Intraoperative total blood loss is the primary endpoint of the trial. Secondary endpoints include blood loss during the hepatectomy, the duration of both the hepatectomy and the entire surgical procedure, as well as blood transfusion requirements of the procedure. To generate reliable data, intraoperative blood loss will be recorded with respect to all rinse fluids during surgery, ascites and by weighing used swabs to generate reliable data. At 80% power and an alpha of 0.025 for both either of the experimental groups, twenty-three subjects will be analysed per protocol in each study arm in order to detect a clinically relevant reduction of intraoperative blood loss. The intention to treat analysis will include sixty-nine patients. The follow up period for each patient will be 90 days for safety reasons, whereas all clinical outcomes will be measured within the first ten postoperative days. This is the first prospective, randomized trial comparing two innovative, technical methods of vessel sealing and dissection against standard techniques for recipient hepatectomy. This will be done to detect a relevant reduction of intraoperative blood loss during liver transplantation.The results of the trial are expected to improve patients' outcome and safety after liver transplantation and to increase the general safety of this procedure.

DETAILED DESCRIPTION:
Liver transplantation (LT) is a well-established procedure for the treatment of end stage liver disease. Many improvements in the surgical technique rendered this operation relatively safe. Most important operative innovations after the initial introduction of LT in the clinical Routine undertaken by Starzl include the use of veno-venous bypass in LT, the piggy-back technique with preservation of the recipients' caval vein and it's modification which was introduced by Belghiti with side-to-side cavo-caval anastomosis. Nevertheless very few improvements have been introduced in the surgical technique with regards to tissue preparation and sealing the blood vessels during recipient hepatectomy. Due to end stage liver disease and both the recipients' general and coagulatory condition, the hepatectomy carries the risk of severe blood loss which can impair the outcome after LT. Usually the recipient hepatectomy is carried out as a combination of sharp dissection of the hepatic adhesions to the abdominal wall and the diaphragm and clip or suture ligature of small retrohepatic caval vein branches.

With advances in surgical procedures and equipment, modern technologies have been introduced, which have shortened operation time and improved surgical outcomes. Exquisite equipment for liver parenchyma transection, such as Cavitron ultrasonic surgical aspirator, ultrasonic dissector (USD), LigaSure (LS) and Tissue Link can also be used to reduce hemorrhage in liver resection. The ultrasonic scalpel (Ethicon) is a new USD that cuts and coagulates tissue using ultrasound at frequencies higher than those used by an ultrasonic aspirator. This device can also serve as a grasper and basically utilizes a blade which oscillates at 55 kHz, thus producing heat and enabling coagulation of vessels. Recently, its use and potential advantages in open liver resection have been demonstrated. The main technical advancement in this field relates to decreased intra-operative bleeding. Results of using USD (Harmonic Scalpel) during recipient hepatectomy showed that this method is safe compared with conventional knot tying ligation regarding intra- and postoperative bleeding rate. The electrothermal bipolar vessel sealing device LS is another alternative, which applies electrothermal bipolar coagulation and dissection in one step. The LS dissection device seals the tissue first before it is divided (both Tasks are performed with the same device). This may prevent severe bleeding. Furthermore, the sealing device is capable of coping with the small liver veins which can be sealed and divided safely without the need for sutures or clips. Especially the latter of which is known for interfering with sufficient "tangential" clamping of the inferior caval vein (IVC) for side to side cavo-cavostomy during piggy-back LT. It was reported that the use of LS devices for recipient hepatectomy in LT. It was concluded that, LS vessel sealing was an efficient method and that vessel sealing of the caval and Portal veins as well as other structures could be safely performed in the setting of end-stage liver disease.

To our knowledge, no randomized clinical trial has been conducted to compare various innovative dissection methods against the standard techniques used for recipient hepatectomy. While LS and USD have been proven to be used safely in several major surgical procedures, including liver resection, their ability to reduce blood loss in liver transplant recipient hepatectomy has not yet been evaluated systematically.

ELIGIBILITY:
Inclusion Criteria:

* Allocation of donor liver via Eurotransplant to recipient
* Recipients must be aged 18 or older
* A signed, written informed consent for participation in the trial

Exclusion Criteria:

* High urgency state of recipient
* Previous liver transplantation
* Combined organ transplantation
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Total Blood loss during surgical procedure | One day
  The suction container fluid volume (in 20 milliliters) will be added to the weight (in grams) of all surgical swabs at the end of skin closure procedures (A). The difference of the density of the rinse solution (isotonic Sodium Chloride solution) and blood is approximately 0.055 g/cm³. Regarding the accuracy of these measurements, this difference is clinically irrelevant.
  The volume of the entire rinse fluid (in milliliters) that is used during the procedure and the amount of ascites (in milliliters) will be added to the known dry weight (in grams) of the respective number of surgical swabs that are used during the procedure and the known dry weight of the drip catching swab container (B).
  The total blood loss is defined as "A" minus "B" in milliliters.

SECONDARY OUTCOMES:
Blood loss during recipient hepatectomy | One day
Time from skin incision to end of hemostasis after hepatectomy | One day
Time from skin incision to end of skin closure | One day
Hemodynamic status during surgery | One day
  Data on the mean arterial pressure and central venous pressure will be obtained at the beginning of hepatectomy after incision and adhesiolysis.
The number of packed red blood cells (PRBC) units transfused during surgery | One day
The number of fresh frozen plasma (FFP) units transfused during surgery | One day
The number of platelet units transfused during surgery | One day
Conversion rate | One day
  Conversion rate to alternative methods during recipient hepatectomy in LS and USD groups
Coagulation state | Ten days
  International Normalized Ratio, partial thromboplastin time and platelet levels of patients will be recorded pre- and postoperatively until POD 10.
Hemoglobin level | Ten days
  Hemoglobin Levels of patients will be recorded pre- and postoperatively until POD 10.
Postoperative PRBC and FFP Transfusion until POD 10 | Ten days
Postoperative bleeding | Ten days
  Postoperative hemorrhaging until POD 10 will be recorded and classified according to the Clavien-Dindo classification.
Postoperative morbidity | Three months
  Postoperative morbidity will be recorded and classified according to the Clavien-Dindo classification.
Retransplantation rate | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Houben, MD, Principal Investigator — Department of General, Visceral and Transplant Surgery, University Hospital Heidelberg, Germany

REFERENCES:
- [Derived] Houben P, Khajeh E, Hinz U, Knebel P, Diener MK, Mehrabi A. SEALIVE: the use of technical vessel-sealing devices for recipient hepatectomy in liver transplantation: study protocol for a randomized controlled trial. Trials. 2018 Jul 16;19(1):380. doi: 10.1186/s13063-018-2778-1. PMID 30012178